CLINICAL TRIAL: NCT04278326
Title: Primary Organoid Models and Combined Nucleic Acids Therapeutics for Innovative Anti-HPV Treatments in Cervico-vaginal Cancers and Precancerous Lesions
Brief Title: Primary Organoid Models and Combined Nucleic Acids Therapeutics for Anti-HPV Treatments
Acronym: ORGANOIDES
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: the partner laboratory encountered various difficulties (COVID, relocation of the laboratory, personnel problems), which prevented the organoid model from being built
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Collaborators: CNRS - Pr Chantal PICHON (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHRO-2019-08
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: HPV Infection; Vaginal Cancer; Cervical Dysplasia; Cervical Cancer
Keywords: vaginal organoid; human papilloma virus; nucleic acids; cervical dysplasia; cervical cancer
MeSH Terms: conditions — Papillomavirus Infections; Vaginal Neoplasms; Uterine Cervical Dysplasia; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): 1. Patients infected by oncogenic HPV and presented a high grade cervical dysplasia or a cervical cancer
  2. Patients with cervical or vaginal cancer
  3. All patients
  Interventions: Procedure: Vaginal Biopsy

INTERVENTIONS:
Procedure: Vaginal Biopsy — 1. Vaginal biopsies
  2. Additional cervical and vaginal biopsies
  3. Non invasive cervico-vaginal swab like a smear

SUMMARY:
Human papilloma virus (HPV) is responsible of the most common sexually transmitted infection. It can cause severe cancer lesions, of the cervix, vulva, vagina, penis and oropharynx. The International Agency for Cancer Research of World Health Organization (WHO) classified a dozen of HPV related high-risk cancer types, and recognized cervical cancer as the most common HPV-related disease. HPV 16 and 18 are responsible for 70% of cervical cancers.

Due to the few symptoms of cervical cancer, women are often diagnosed with advanced state. Current treatments imply cervical conisation or hysterectomy, with or without lymphadenectomy and or radiotherapy, or chemotherapy.

However, few pharmacological options are available against oncogenic papilloma viruses and thus against recurrences The aim of this project is to develop relevant organoids models from patient biopsies that will be used to identify biomarkers and evaluate in a closest preclinical setting novel nucleic acids based therapeutic strategy for HPV-cervical-vaginal dysplasia and cancers.

DETAILED DESCRIPTION:
In this project, the investigators want to develop organotypic culture of primary-derived biopsies, and combine them with organ-on-a-chip technology, to better characterize the HPV infection and cancer progression, as well as to screen innovative treatments for cervical and vaginal cancers.

Our study will cover cervical dysplasia and cervical cancers HPV induced. The investigators will perform cervical and or vaginal biopsies from patients with oncogenic HPV lesions. A protocol validated to collect biopsies from precancerous cervico-vaginal lesions or cervical cancer patients in CHRO (Orleans, France). The biopsies will be performed during a consultation in the Hospital center of Orleans, or in the theatre room during a conisation or an hysterectomy. The PRIMMO platform is the research platform of Regional hospital center of Orleans (CHRO) dedicated to the promotion of translational research. It will be involved in the collection, analysis and biobank storage setup of the project. Fresh samples will be collected and bring directly to the lab for organoid cell culture development. Detection of HPV in each biopsy will be carried out by the PRIMMO platform.

The organoid development from patient biopsies will take place into the lab of the Biophysic Molecular center in Orleans.

The organoids will be selected according to three criteria: their ability to grow until a first passage, their doubling time and their ability to be frozen and resuscitated. Such organoids maintain pathogen-host interaction and better model physiopathology of vaginal cervical dysplasia CIN2-3 or cervical cancer and thus allow for the detection of biomarkers for pre-cancerous lesions. In addition, organoids reduce the use of animal models and can be used for drug screening, In a second step, the investigators propose to use mRNA to produce in situ the nanobodies targeting E6 and E7, to inhibit viral replication and tumor growth

Socio-epidemiological data will be collected for each patient, in the form of a table.

The study could be stopped in case of serious undesirable events. Safety evaluation As this is a category 2 study, no particular vigilance linked to the research protocol will be useful.

However, the monitoring and reporting of unexpected events resulting from participation in the study will be declared to the "materiovigilance site" of the CHR of Orleans Given the minimal risks associated with the study, an independent monitoring committee was not considered necessary.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 75 years old.
* Patients presented with cervical or vaginal dysplasia or cancer induced by oncogenic HPV demonstrated by a PAP test and or HPV testing requiring a biopsy and histology in current care.

Patients with previous history of conisation or hysterectomy for lesions of the cervix or the vagina caused by oncogenic HPV.

To participate in the study, patients must sign an informed consent.

Exclusion Criteria:

* - Pregnant women
* Patients with coagulation disorders
* Refusal of patients to participate in the trial Patients not affiliated to medical insurance
* Person deprived of their liberty by judicial or administrative decision
* Adults over 18 who are under legal protection measures or cannot give their consent

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
To develop a 3D vaginal organoid culture model. | 4 years
  The main objective is to develop a 3D cell culture model of organoid type from vaginal and cervical biopsies of patients infected with an oncogenic papilloma virus

SECONDARY OUTCOMES:
Inhibition of HPV molecular therapeutics using oligonucleotide, and siRNA (small interfering RNA) | 4 years
  To be able to use a vaginal cellular 3D model to develop an anti-HPV treatment

CONTACTS AND LOCATIONS:
Overall Officials: Souhail ALOUINI, M.D.,Ph.D., Principal Investigator — CHR Orléans; Chantal PICHON, Ph.D., Study Chair — Centre National de la Recherche Scientifique, France
Locations (1):
- CHR Orléans, Orléans, France

REFERENCES:
- [Background] Ngamkham J, Boonmark K, Phansri T. Detection and Type-Distribution of Human Papillomavirus in Vulva and Vaginal Abnormal Cytology Lesions and Cancer Tissues from Thai Women. Asian Pac J Cancer Prev. 2016;17(3):1129-34. doi: 10.7314/apjcp.2016.17.3.1129. PMID 27039737
- [Background] Duke P, Godwin M, Ratnam S, Dawson L, Fontaine D, Lear A, Traverso-Yepez M, Graham W, Ravalia M, Mugford G, Pike A, Fortier J, Peach M. Effect of vaginal self-sampling on cervical cancer screening rates: a community-based study in Newfoundland. BMC Womens Health. 2015 Jun 10;15:47. doi: 10.1186/s12905-015-0206-1. PMID 26060041
- [Background] Koo YJ, Min KJ, Hong JH, Lee JK. Efficacy of Poly-Gamma-Glutamic Acid in Women with High-Risk Human Papillomavirus-Positive Vaginal Intraepithelial Neoplasia: an Observational Pilot Study. J Microbiol Biotechnol. 2015 Jul;25(7):1163-9. doi: 10.4014/jmb.1503.03106. PMID 25907060
- [Background] Mollers M, King AJ, Knol MJ, Scherpenisse M, Meijer CJ, van der Klis FR, de Melker HE. Effectiveness of human papillomavirus vaccine against incident and persistent infections among young girls: Results from a longitudinal Dutch cohort study. Vaccine. 2015 May 28;33(23):2678-83. doi: 10.1016/j.vaccine.2015.04.016. Epub 2015 Apr 14. PMID 25887090
- [Background] Wang KD, Xu DJ, Wang BY, Yan DH, Lv Z, Su JR. Inhibitory Effect of Vaginal Lactobacillus Supernatants on Cervical Cancer Cells. Probiotics Antimicrob Proteins. 2018 Jun;10(2):236-242. doi: 10.1007/s12602-017-9339-x. PMID 29071554